CLINICAL TRIAL: NCT03861390
Title: Phase I/II Randomized, Double-blind, Placebo-controlled Cross-over Study of Prednisone on Airway Inflammatory Response to Inhaled Wood Smoke
Brief Title: Woodsmoke Particulate + Prednisone
Acronym: Smokisone
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 18-2196
Record Dates: First submitted 2019-03-01; First posted 2019-03-04 (Actual); Results first posted 2024-05-23 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-04

CONDITIONS: Airway Inflammation
MeSH Terms: interventions — Prednisone

STUDY DESIGN:
Intervention Model Description: The randomization schedule will be generated by using permuted block randomization with a block size of 4 (2 prednisone, 2 placebo for the first treatment period of the protocol).
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prednisone, then Placebo (Active Comparator): Participants will receive prednisone following WSP exposure. After a 4-week washout period, participants will receive placebo following WSP exposure.
  Interventions: Drug: 60 mg Prednisone; Drug: Placebo
- Placebo, then Prednisone (Placebo Comparator): Participants will receive placebo following WSP exposure. After a 4-week washout period, participants will receive prednisone following WSP exposure.
  Interventions: Drug: 60 mg Prednisone; Drug: Placebo

INTERVENTIONS:
Drug: 60 mg Prednisone — Immediately following exit from the wood smoke chamber, subjects will receive 60 mg of prednisone per randomization schema
Drug: Placebo — Immediately following exit from the wood smoke chamber, subjects will receive a matching placebo to the 60 mg of prednisone per randomization schema

SUMMARY:
Deployment of military personnel has been associated with increased respiratory illness likely due, in part, to inhalation of unusual particulate matter (PM), such as from burn pits. Inflammation is a key initial response to inhaled particulates. The researchers have developed a protocol using inhaled wood smoke particles (WSP) as a way to study PM-induced airway inflammation. Exposure to wood smoke particles causes symptoms, even in healthy people, such as eye irritation, cough, shortness of breath, and increased mucous production. The purpose of this research study is to see if an oral steroid treatment can reduce the airway inflammation caused by the inhaled WSP. The exposure will be 500 µg/m³ of WSP for 2 hours, with intermittent exercise on a bicycle and rest. The wood is burned in a typical wood stove and piped into the chamber.

DETAILED DESCRIPTION:
Military deployment is associated with exposure to novel particulate matter (PM), such as from burn pits, aeroallergens, and increased cigarette consumption. War fighters exposed to these inhalational exposures exhibit immediate and chronic respiratory morbidity. For example, military service personnel surveyed in both the Republic of Korea (ROK) and Kabul, Afghanistan reported a general increase in respiratory morbidity, including asthma and chronic bronchitis, associated with their deployment. Air contaminants in the ROK were characterized by elevated levels of both PM 0.5-2.5 and PM 2.5-10. Similarly, exposures in Kabul were characterized by multiple airborne PM exposures, including those from burn pits. Burn pit PM includes metals, bioaerosols, organic by-products, and biomass combustion particles. These findings indicate that inhaled PM is a likely cause of respiratory morbidity in the field.

Inflammation is a key initial response to inhaled particulates. Wood smoke particles (WSP) serve as a model agent to study PM-induced bronchitis. WSP inhalation generates reactive oxidant (and nitrosative) species which cause local injury of airway epithelial cells and release of damage-associated molecular patterns (DAMPs) that activate toll-like receptors (TLR) and Interleukin (IL)-1-mediated innate immune responses by resident airway macrophages. Contamination of PM with bioaerosols, which contain lipopolysaccharide (LPS), also activates innate immune responses through toll-like receptor 4 (TLR4) activation of resident airway macrophages. These complementary processes result in recruitment of neutrophils (PMN), which mediate luminal airway inflammation with release of toxic mediators such as neutrophil elastase and myeloperoxidase that promote acute and chronic bronchitis.

Therefore, mitigation of PM-induced airway neutrophilic inflammation should be a key focus in order to reduce the respiratory morbidity of military personnel. The researchers have studied a number of pro-inflammatory inhaled agents, such as nebulized LPS, ozone (O3), and WSP, as models of acute neutrophilic bronchitis against which to test a number of therapeutic agents. To this effect, the researchers have reported that inhaled fluticasone inhibits O3-induced and LPS-induced neutrophilic inflammation, and that parenteral anakinra and oral gamma-tocopherol inhibit neutrophilic responses to inhaled LPS. In this study, the researchers will evaluate the efficacy of oral prednisone, a readily available anti-inflammatory medication commonly used in airway inflammatory diseases, in mitigating WSP-induced airway inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45 years, inclusive, of both genders
* Negative pregnancy test for females who are not s/p hysterectomy with oophorectomy
* No history of episodic wheezing, chest tightness, or shortness of breath consistent with asthma, or physician-diagnosed asthma.
* Forced expiratory volume at one second (FEV1) of at least 80% of predicted and FEV1/ forced vital capacity (FVC) ≥0.70.
* Oxygen saturation of ≥93%
* Ability to provide an induced sputum sample.
* Subject must demonstrate a ≥10% increase in sputum %PMNs 6 hours following inhaled WSP exposure, when compared to baseline sputum (to be completed in a separate protocol # 15-1775).
* Proof of vaccination to COVID-19.

Exclusion Criteria:

Clinical contraindications:

* Any chronic medical condition considered by the PI as a contraindication to the exposure study including significant cardiovascular disease, diabetes, chronic renal disease, chronic thyroid disease, history of chronic infections/immunodeficiency.
* Viral upper respiratory tract infection within 4 weeks of challenge.
* Any acute infection requiring antibiotics within 4 weeks of exposure or fever of unknown origin within 4 weeks of challenge.
* Abnormal physical findings at the baseline visit, including but not limited to abnormalities on auscultation, temperature of 37.8° C, Systolic BP > 150mm Hg or < 85 mm Hg; or Diastolic BP > 90 mm Hg or < 50 mm Hg, or pulse oximetry saturation reading less than 93%.
* Physician diagnosis of asthma
* If there is a history of allergic rhinitis, subjects must be asymptomatic of allergic rhinitis at the time of study enrollment.
* Mental illness or history of drug or alcohol abuse that, in the opinion of the investigator, would interfere with the participant's ability to comply with study requirements.
* Medications which may impact the results of the WSP exposure, interfere with any other medications potentially used in the study (to include steroids, beta antagonists, non-steroidal anti-inflammatory agents)
* Cigarette smoking > 1 pack per month
* Unwillingness to use reliable contraception if sexually active (IUD, birth control pills/patch, condoms).
* Use of immunosuppressive or anticoagulant medications including routine use of NSAIDS. Oral contraceptives are acceptable, as are antidepressants and other medications may be permitted if, in the opinion of the investigator, the medication will not interfere with the study procedures or compromise safety and if the dosage has been stable for 1 month.
* Orthopedic injuries or impediments that would preclude bicycle or treadmill exercise.
* Inability to avoid NSAIDS, Multivitamins, Vitamin C or E or herbal supplements.
* Allergy/sensitivity to study drugs or their formulations
* Positive COVID-19 test in the past 90 days
* Pregnant/lactating women and children (< 18 years as this is age of majority in North Carolina) will also be excluded since the risks associated with WSP exposure to the fetus or child, respectively, are unknown and cannot be justified for this non-therapeutic protocol. Individuals over 45 years of age will not be included due to the increased possibility of co-morbidities and need for prohibited medications.
* Inability or unwillingness of a participant to give written informed consent

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2019-03-22 (Actual); Primary Completion 2023-05-12 (Actual); Study Completion 2023-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terry Noah, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Center for Environmental Medicine, Asthma and Lung Biology at UNC Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pugh MJ, Jaramillo CA, Leung KW, Faverio P, Fleming N, Mortensen E, Amuan ME, Wang CP, Eapen B, Restrepo M, Morris MJ. Increasing Prevalence of Chronic Lung Disease in Veterans of the Wars in Iraq and Afghanistan. Mil Med. 2016 May;181(5):476-81. doi: 10.7205/MILMED-D-15-00035. PMID 27136656
- [Background] Korzeniewski K, Nitsch-Osuch A, Konior M, Lass A. Respiratory tract infections in the military environment. Respir Physiol Neurobiol. 2015 Apr;209:76-80. doi: 10.1016/j.resp.2014.09.016. Epub 2014 Sep 30. PMID 25278277
- [Background] Baird CP. Review of the Institute of Medicine report: long-term health consequences of exposure to burn pits in Iraq and Afghanistan. US Army Med Dep J. 2012 Jul-Sep:43-7. No abstract available. PMID 22815164
- [Background] Gomez JC, Yamada M, Martin JR, Dang H, Brickey WJ, Bergmeier W, Dinauer MC, Doerschuk CM. Mechanisms of interferon-gamma production by neutrophils and its function during Streptococcus pneumoniae pneumonia. Am J Respir Cell Mol Biol. 2015 Mar;52(3):349-64. doi: 10.1165/rcmb.2013-0316OC. PMID 25100610
- [Background] Barth SK, Dursa EK, Bossarte R, Schneiderman A. Lifetime Prevalence of Respiratory Diseases and Exposures Among Veterans of Operation Enduring Freedom and Operation Iraqi Freedom Veterans: Results From the National Health Study for a New Generation of U.S. Veterans. J Occup Environ Med. 2016 Dec;58(12):1175-1180. doi: 10.1097/JOM.0000000000000885. PMID 27930474
- [Background] Szema AM. Occupational Lung Diseases among Soldiers Deployed to Iraq and Afghanistan. Occup Med Health Aff. 2013;1:10.4172/2329-6879.1000117. doi: 10.4172/2329-6879.1000117. PMID 24443711
- [Background] Morris MJ, Lucero PF, Zanders TB, Zacher LL. Diagnosis and management of chronic lung disease in deployed military personnel. Ther Adv Respir Dis. 2013 Aug;7(4):235-45. doi: 10.1177/1753465813481022. Epub 2013 Mar 7. PMID 23470637
- [Background] Auerbach A, Hernandez ML. The effect of environmental oxidative stress on airway inflammation. Curr Opin Allergy Clin Immunol. 2012 Apr;12(2):133-9. doi: 10.1097/ACI.0b013e32835113d6. PMID 22306553
- [Background] Alexis NE, Brickey WJ, Lay JC, Wang Y, Roubey RA, Ting JP, Peden DB. Development of an inhaled endotoxin challenge protocol for characterizing evoked cell surface phenotype and genomic responses of airway cells in allergic individuals. Ann Allergy Asthma Immunol. 2008 Mar;100(3):206-15. doi: 10.1016/S1081-1206(10)60444-9. PMID 18426139
- [Background] Hernandez ML, Harris B, Lay JC, Bromberg PA, Diaz-Sanchez D, Devlin RB, Kleeberger SR, Alexis NE, Peden DB. Comparative airway inflammatory response of normal volunteers to ozone and lipopolysaccharide challenge. Inhal Toxicol. 2010 Jul;22(8):648-56. doi: 10.3109/08958371003610966. PMID 20540623
- [Background] Hernandez M, Brickey WJ, Alexis NE, Fry RC, Rager JE, Zhou B, Ting JP, Zhou H, Peden DB. Airway cells from atopic asthmatic patients exposed to ozone display an enhanced innate immune gene profile. J Allergy Clin Immunol. 2012 Jan;129(1):259-61.e1-2. doi: 10.1016/j.jaci.2011.11.007. PMID 22196529
- [Background] Alexis NE, Peden DB. Blunting airway eosinophilic inflammation results in a decreased airway neutrophil response to inhaled LPS in patients with atopic asthma: a role for CD14. J Allergy Clin Immunol. 2001 Oct;108(4):577-80. doi: 10.1067/mai.2001.118511. PMID 11590384
- [Background] Hernandez ML, Mills K, Almond M, Todoric K, Aleman MM, Zhang H, Zhou H, Peden DB. IL-1 receptor antagonist reduces endotoxin-induced airway inflammation in healthy volunteers. J Allergy Clin Immunol. 2015 Feb;135(2):379-85. doi: 10.1016/j.jaci.2014.07.039. Epub 2014 Sep 5. PMID 25195169
- [Background] Hernandez ML, Wagner JG, Kala A, Mills K, Wells HB, Alexis NE, Lay JC, Jiang Q, Zhang H, Zhou H, Peden DB. Vitamin E, gamma-tocopherol, reduces airway neutrophil recruitment after inhaled endotoxin challenge in rats and in healthy volunteers. Free Radic Biol Med. 2013 Jul;60:56-62. doi: 10.1016/j.freeradbiomed.2013.02.001. Epub 2013 Feb 9. PMID 23402870
- [Background] Burbank AJ, Duran CG, Pan Y, Burns P, Jones S, Jiang Q, Yang C, Jenkins S, Wells H, Alexis N, Kesimer M, Bennett WD, Zhou H, Peden DB, Hernandez ML. Gamma tocopherol-enriched supplement reduces sputum eosinophilia and endotoxin-induced sputum neutrophilia in volunteers with asthma. J Allergy Clin Immunol. 2018 Apr;141(4):1231-1238.e1. doi: 10.1016/j.jaci.2017.06.029. Epub 2017 Jul 20. PMID 28736267
- [Background] National Asthma Education and Prevention Program. Expert Panel Report 3 (EPR-3): Guidelines for the Diagnosis and Management of Asthma-Summary Report 2007. J Allergy Clin Immunol. 2007 Nov;120(5 Suppl):S94-138. doi: 10.1016/j.jaci.2007.09.043. PMID 17983880
- [Background] Walters JA, Tan DJ, White CJ, Wood-Baker R. Different durations of corticosteroid therapy for exacerbations of chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2018 Mar 19;3(3):CD006897. doi: 10.1002/14651858.CD006897.pub4. PMID 29553157
- [Background] Stern A, Skalsky K, Avni T, Carrara E, Leibovici L, Paul M. Corticosteroids for pneumonia. Cochrane Database Syst Rev. 2017 Dec 13;12(12):CD007720. doi: 10.1002/14651858.CD007720.pub3. PMID 29236286
- [Background] Venekamp RP, Thompson MJ, Hayward G, Heneghan CJ, Del Mar CB, Perera R, Glasziou PP, Rovers MM. Systemic corticosteroids for acute sinusitis. Cochrane Database Syst Rev. 2014 Mar 25;2014(3):CD008115. doi: 10.1002/14651858.CD008115.pub3. PMID 24664368
- [Background] Ghio AJ, Soukup JM, Case M, Dailey LA, Richards J, Berntsen J, Devlin RB, Stone S, Rappold A. Exposure to wood smoke particles produces inflammation in healthy volunteers. Occup Environ Med. 2012 Mar;69(3):170-5. doi: 10.1136/oem.2011.065276. Epub 2011 Jun 30. PMID 21719562
- [Background] Esther CR Jr, Lazaar AL, Bordonali E, Qaqish B, Boucher RC. Elevated airway purines in COPD. Chest. 2011 Oct;140(4):954-960. doi: 10.1378/chest.10-2471. Epub 2011 Mar 31. PMID 21454402
- [Background] Jones B, and Kenward, M.G. . Design and analysis of cross-over trials. Third ed: CRC Press; 2015
- [Background] Alexis NE, Zhou H, Lay JC, Harris B, Hernandez ML, Lu TS, Bromberg PA, Diaz-Sanchez D, Devlin RB, Kleeberger SR, Peden DB. The glutathione-S-transferase Mu 1 null genotype modulates ozone-induced airway inflammation in human subjects. J Allergy Clin Immunol. 2009 Dec;124(6):1222-1228.e5. doi: 10.1016/j.jaci.2009.07.036. PMID 19796798

RESULTS

PARTICIPANT FLOW:
Groups:
- Prednisone, Then Placebo: Participants will receive prednisone following wood smoke particle (WSP) exposure. After a 4-week washout period, participants will receive placebo following WSP exposure.
  60 mg Prednisone: Immediately following exit from the wood smoke chamber, subjects will receive 60 mg of prednisone per randomization schema
  Placebo: Immediately following exit from the wood smoke chamber, subjects will receive a matching placebo to the 60 mg of prednisone per randomization schema
- Placebo, Then Prednisone: Participants will receive placebo following wood smoke particle (WSP) exposure. After a 4-week washout period, participants will receive prednisone following WSP exposure.
  60 mg Prednisone: Immediately following exit from the wood smoke chamber, subjects will receive 60 mg of prednisone per randomization schema
  Placebo: Immediately following exit from the wood smoke chamber, subjects will receive a matching placebo to the 60 mg of prednisone per randomization schema
Period: First Intervention
Arm/Group | Prednisone, Then Placebo | Placebo, Then Prednisone
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: Washout (4 Weeks)
Arm/Group | Prednisone, Then Placebo | Placebo, Then Prednisone
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: Period Title: Second Intervention
Arm/Group | Prednisone, Then Placebo | Placebo, Then Prednisone
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Prednisone, Then Placebo: Participants receive prednisone following WSP exposure. After a 4-week washout period, participants receive placebo following WSP exposure.
  60 mg Prednisone: Immediately following exit from the wood smoke chamber, subjects receive 60 mg of prednisone per randomization schema
  Placebo: Immediately following exit from the wood smoke chamber, subjects receive a matching placebo to the 60 mg of prednisone per randomization schema
- Placebo, Then Prednisone: Participants receive placebo following WSP exposure. After a 4-week washout period, participants receive prednisone following WSP exposure.
  60 mg Prednisone: Immediately following exit from the wood smoke chamber, subjects receive 60 mg of prednisone per randomization schema
  Placebo: Immediately following exit from the wood smoke chamber, subjects receive a matching placebo to the 60 mg of prednisone per randomization schema
- Total: Total of all reporting groups
Arm/Group | Prednisone, Then Placebo | Placebo, Then Prednisone | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 12
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 3 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 6 | 5 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 5 | 4 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 4 Hours in Sputum Percent Neutrophils
Description: Change in sputum percent neutrophils from baseline to 4 hours post WSP exposure
Time Frame: Baseline, 4 hours post WSP exposure
Population: Cell differential slide inadequate for 1 participant in prednisone arm; paired analysis drops this participant from analysis across both arms.
Measure: Median (Inter-Quartile Range); unit: percent neutrophils
Groups:
- Prednisone: Immediately following exit from the wood smoke chamber, subjects receive 60 mg of prednisone per randomization schema
- Placebo: Immediately following exit from the wood smoke chamber, subjects receive a matching placebo to the 60 mg of prednisone per randomization schema
Arm/Group | Prednisone | Placebo
Number analyzed (Participants) | 11 | 11
percent neutrophils | -2.62 [-6.27 to 6.08] | 5.45 [1.21 to 8.79]
Statistical Analysis 1: Comparison: Prednisone vs Placebo; Test type: Other; p = 0.24, Wilcoxon (Mann-Whitney) — The a priori threshold for statistical significance is < 0.05

2. Primary Outcome: Change From Baseline to 24 Hours in Sputum Percent Neutrophils
Description: Change in sputum percent neutrophils from baseline to 24 hours post WSP exposure
Time Frame: Baseline, 24 hours post WSP exposure
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percent neutrophils
Arm/Group | Prednisone | Placebo
Number analyzed (Participants) | 11 | 11
percent neutrophils | 8.07 [-0.34 to 26.00] | 22.68 [7.00 to 41.40]
Statistical Analysis 1: Comparison: Prednisone vs Placebo; Test type: Other; p = 0.17, Wilcoxon (Mann-Whitney) — The a priori threshold for statistical significance is < 0.05

3. Secondary Outcome: Change in Number of Sputum Neutrophils
Description: Neutrophil numbers/mg measured at 4 and 24 hours post WSP exposure. Comparisons at 4 and 24 hours are each made with respect to Baseline.
Time Frame: Baseline, 4 and 24 hours post WSP exposure
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Neutrophils/mg
Arm/Group | Prednisone | Placebo
Number analyzed (Participants) | 11 | 11
Neutrophils/mg
  4 hours post WSP exposure | 52.00 [-120.00 to 76.00] | 36.00 [-6.00 to 73.00]
  24 hours post WSP exposure | -17.00 [-53.00 to 92.00] | 37.00 [-13.00 to 143.00]
Statistical Analysis 1: Comparison: Prednisone vs Placebo; 4 hours post WSP exposure; Test type: Other; p = 0.70, Wilcoxon (Mann-Whitney) — The a priori threshold for statistical significance is < 0.05
Statistical Analysis 2: Comparison: Prednisone vs Placebo; 24 hours post WSP exposure; Test type: Other; p = 0.37, Wilcoxon (Mann-Whitney) — The a priori threshold for statistical significance is < 0.05

4. Secondary Outcome: Change in Number of Sputum Eosinophils
Description: Eosinophil numbers/mg measured at 4 and 24 hours post WSP exposure. Comparisons at 4 and 24 hours are each made with respect to Baseline.
Time Frame: Baseline, 4 and 24 hours post WSP exposure
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Eosinophils/mg
Arm/Group | Prednisone | Placebo
Number analyzed (Participants) | 11 | 11
Eosinophils/mg
  4 hours post WSP exposure | 0.00 [-0.5 to 2.00] | 0.00 [0.00 to 0.00]
  24 hours post WSP exposure | 0.00 [-1.00 to 0.00] | 0.00 [0.00 to 1.00]
Statistical Analysis 1: Comparison: Prednisone vs Placebo; 4 hours post WSP exposure; Test type: Other; p = 0.77, Wilcoxon (Mann-Whitney) — The a priori threshold for statistical significance is < 0.05
Statistical Analysis 2: Comparison: Prednisone vs Placebo; 24 hours post WSP exposure; Test type: Other; p = 0.48, Wilcoxon (Mann-Whitney) — The a priori threshold for statistical significance is < 0.05

5. Secondary Outcome: Change in Percent Sputum Eosinophils
Description: Percent eosinophil measured at 4 and 24 hours post WSP exposure. Comparisons at 4 and 24 hours are each made with respect to Baseline.
Time Frame: Baseline, 4 and 24 hours post WSP exposure
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percent eosinophils
Arm/Group | Prednisone | Placebo
Number analyzed (Participants) | 11 | 11
percent eosinophils
  4 hours post WSP exposure | 0.00 [0.00 to 0.00] | 0.00 [-0.20 to 0.30]
  24 hours post WSP exposure | 0.00 [0.00 to 0.00] | 0.00 [-0.20 to 0.20]
Statistical Analysis 1: Comparison: Prednisone vs Placebo; 4 hours post WSP exposure; Test type: Other; p = 0.96, Wilcoxon (Mann-Whitney) — The a priori threshold for statistical significance is < 0.05
Statistical Analysis 2: Comparison: Prednisone vs Placebo; 24 hours post WSP exposure; Test type: Other; p = 0.91, Wilcoxon (Mann-Whitney) — The a priori threshold for statistical significance is < 0.05

6. Secondary Outcome: Change in IL-1b
Description: Interleukin beta (IL-1b) via Mesoscale platform (pg/mL) at 4 and 24 hours post WSP exposure. Comparisons at 4 and 24 hours are each made with respect to Baseline.
Time Frame: Baseline, 4 and 24 hours post WSP exposure
Population: An attempt was made to analyze samples for 12 participants; although some samples had insufficient quantity remaining. Data are reported for all samples that yielded data for each endpoint and at each time.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Prednisone | Placebo
Number analyzed (Participants) | 12 | 12
pg/mL
  4 hours post WSP exposure: number analyzed (Participants) | 12 | 8
  4 hours post WSP exposure | 39.60 [-124.00 to 194.00] | -41.80 [-634.00 to 148.00]
  24 hours post WSP exposure: number analyzed (Participants) | 10 | 9
  24 hours post WSP exposure | 357.00 [16.60 to 546.00] | 128.00 [-461.00 to 197.00]
Statistical Analysis 1: Comparison: Prednisone vs Placebo; 4 hours post WSP exposure; Test type: Other; p = 0.46, Wilcoxon (Mann-Whitney) — The a priori threshold for statistical significance is < 0.05
Statistical Analysis 2: Comparison: Prednisone vs Placebo; 24 hours post WSP exposure; Test type: Other; p = 0.46, Wilcoxon (Mann-Whitney) — The a priori threshold for statistical significance is < 0.05

7. Secondary Outcome: Change in IL-6
Description: Interleukin-6 (IL-6) via Mesoscale platform (pg/mL) at 4 and 24 hours post WSP exposure. Comparisons at 4 and 24 hours are each made with respect to Baseline.
Time Frame: Baseline, 4 and 24 hours post WSP exposure
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Prednisone | Placebo
Number analyzed (Participants) | 12 | 12
pg/mL
  4 hours post WSP exposure: number analyzed (Participants) | 11 | 10
  4 hours post WSP exposure | 52.78 [-310.40 to 231.20] | 80.35 [-131.30 to 472.00]
  24 hours post WSP exposure: number analyzed (Participants) | 11 | 11
  24 hours post WSP exposure | 37.69 [-123.00 to 509.00] | 0.00 [-494.60 to 194.10]
Statistical Analysis 1: Comparison: Prednisone vs Placebo; 4 hours post WSP exposure; Test type: Other; p = 0.82, Wilcoxon (Mann-Whitney) — The a priori threshold for statistical significance is < 0.05
Statistical Analysis 2: Comparison: Prednisone vs Placebo; 24 hours post WSP exposure; Test type: Other — The a priori threshold for statistical significance is < 0.05; p = 0.99, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Change in IL-8
Description: Interleukin-8 (IL-8) via Mesoscale platform (pg/mL) at 4 and 24 hours post WSP exposure. Comparisons at 4 and 24 hours are each made with respect to Baseline.
Time Frame: Baseline, 4 and 24 hours post WSP exposure
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Prednisone | Placebo
Number analyzed (Participants) | 12 | 12
pg/mL
  4 hours post WSP exposure: number analyzed (Participants) | 11 | 9
  4 hours post WSP exposure | 1416.00 [-2161.00 to 7096.00] | 869.00 [-11445.00 to 3866.00]
  24 hours post WSP exposure: number analyzed (Participants) | 10 | 10
  24 hours post WSP exposure | 4835.00 [-2007.00 to 17149.00] | 627.00 [-6788.00 to 8724.00]
Statistical Analysis 1: Comparison: Prednisone vs Placebo; 4 hours post WSP exposure; Test type: Other; p = 0.38, Wilcoxon (Mann-Whitney) — The a priori threshold for statistical significance is < 0.05
Statistical Analysis 2: Comparison: Prednisone vs Placebo; 24 hours post WSP exposure; Test type: Other; p = 0.84, Wilcoxon (Mann-Whitney) — The a priori threshold for statistical significance is < 0.05

9. Secondary Outcome: Change in TNFa
Description: Tumor necrosis factor alpha (TNFa) via Mesoscale platform (pg/mL) at 4 and 24 hours post WSP exposure. Comparisons at 4 and 24 hours are each made with respect to Baseline.
Time Frame: Baseline, 4 and 24 hours post WSP exposure
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Prednisone | Placebo
Number analyzed (Participants) | 12 | 12
pg/mL
  4 hours post WSP exposure: number analyzed (Participants) | 10 | 11
  4 hours post WSP exposure | -3.63 [-85.50 to 3.45] | 0.00 [-119.00 to 265.00]
  24 hours post WSP exposure: number analyzed (Participants) | 11 | 11
  24 hours post WSP exposure | 17.70 [-17.80 to 115.00] | 0.00 [-237.00 to 73.10]
Statistical Analysis 1: Comparison: Prednisone vs Placebo; 4 hours post WSP exposure; Test type: Other; p = 0.49, Wilcoxon (Mann-Whitney) — The a priori threshold for statistical significance is < 0.05
Statistical Analysis 2: Comparison: Prednisone vs Placebo; 24 hours post WSP exposure; Test type: Other; p = 0.52, Wilcoxon (Mann-Whitney) — The a priori threshold for statistical significance is < 0.05

10. Other Pre Specified Outcome: Mucociliary Clearance (MCC)
Description: 4 hours post WSP exposure, the MCC is done. A whole lung region of interest (ROI) bordering the right lung is used to estimate (by computer analysis) whole lung retention of inhaled radiolabeled particles. Labeled particle counts are measured over a 2 hour period to determine the fraction of initial particle counts remaining. From this data, the investigators will determine the percentage of labeled particles cleared from the lung during the 2 hour observation period.
Time Frame: 4 hours post WSP exposure
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From the time of signing informed consent through study completion, approximately 3 months.
Arm/Group | Prednisone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 5/12 | 4/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prednisone (N=12) | Placebo (N=12)
Bed bug infestation (Social circumstances) | 1 (1) | 0 (0)
Sweating (General disorders) | 1 (2) | 2 (5)
Runny nose (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Eye irritation (Eye disorders) | 1 (1) | 1 (1)
Headache (General disorders) | 1 (1) | 1 (1)
Dry throat (General disorders) | 3 (6) | 1 (1)
Sore throat (General disorders) | 3 (6) | 1 (1)
Drop in FEV1 following sputum induction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
High heart rate alarm (Cardiac disorders) | 0 (0) | 1 (1) — Heart rate exceeded 75 percent of maximum heart rate
Irritation of the nose (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Stuffy nose (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-23): https://cdn.clinicaltrials.gov/large-docs/90/NCT03861390/Prot_SAP_000.pdf